CLINICAL TRIAL: NCT00358969
Title: Guanfacine in the Treatment of Borderline Personality Disorder
Brief Title: Guanfacine to Treat Borderline Personality Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Organization: Bronx VA Medical Center (U.S. Federal Agency)
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GCO 06-0518
Record Dates: First submitted 2006-07-31; First posted 2006-08-01 (Estimated); Last update posted 2006-08-01 (Estimated); Status verified 2006-07

CONDITIONS: Borderline Personality Disorder
Keywords: borderline personality disorder; guanfacine; impulsivity; aggression; affective instability
MeSH Terms: conditions — Borderline Personality Disorder; Impulsive Behavior; Aggression | interventions — Guanfacine

INTERVENTIONS:
Drug: guanfacine (Tenex)

SUMMARY:
This study is designed to investigate whether guanfacine (Tenex) is an effective treatment for borderline personality disorder (BPD), an illness often characterized by unstable mood and impulsive aggression. Guanfacine stimulates activity in the front portion of the brain, a region associated with attention and the control of behavior. We believe that guanfacine may improve symptoms of BPD by improving attention and aiding regulation of behavior.

DETAILED DESCRIPTION:
This is an 8-week treatment study designed to test whether guanfacine is an effective treatment for borderline personality disorder (BPD). Prior to taking the study medication, subjects will have medical and psychiatric evaluations, complete self-report questionnaires, do a functional MRI scan, and complete a set of cognitive tests. While taking the study medication, participants will meet weekly with a study doctor and be administered interviews and questionnaires. At the end of the 8-week trial, participants will be asked to repeat the MRI scan and cognitive tests.

ELIGIBILITY:
Inclusion Criteria: This study includes men and women between the ages of 18 and 55 who meet criteria for borderline personality disorder with impulsive aggression.

Exclusion Criteria: Subjects must not currently be taking any psychiatric medications. Subjects must not meet criteria for current substance dependence, current major depression, bipolar disorder, or schizophrenia-spectrum disorders.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Dates: Start 2006-07

PRIMARY OUTCOMES:
measures of impulsive aggression
measures of affective disturbance
measures of social and occupational functioning
measures of overall clinical status

CONTACTS AND LOCATIONS:
Overall Officials: Antonia S. New, M.D., Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai Hospital - Mood & Personality Research Group, New York, New York, United States